## <u>Project Title</u>: A Telerehabilitation Approach to Enhance Quality of Life Through Exercise Among Adults With Paraplegia: Study Protocol.

NCT number: NCT02833935

## **Principal Investigator**

Shane Sweet, Ph.D.

Department of Kinesiology & Physical Education, Faculty of Education, McGill University Telephone: (514) 398-4184 ext. 09903 Email: shane.sweet@mcgill.ca

## **Statistical Analyses**

Due to pilot nature of this intervention, several approaches were performed to provide a comprehensive examination of the data. First, Hedges' g effect sizes were computed, comparing the intervention to the control group at both six and 10 weeks for each variable. Data were entered into an effect size calculator to provide a Hedge's g with 95% confidence intervals. When large between group differences were found, a measure of effect size, dppc, for mean differences of groups with unequal sample size within a pre-post-control design (Morris, 2008) was calculated. All effect sizes were obtained using the calculator found on www.psychometrica.de/effect size.html#cohenb. A Hedge's g of 0.2, 0.5 and 0.8 represented a small, moderate and large effect size, respectively (Lakens, 2013). These same cut points were used to interpret dppc. Reliable change indices were calculated for the primary outcomes and LTPA. Using the means and standard deviations at baseline, 6, and 10 weeks, and the Cronbach's alpha at baseline, reliable change indices were estimates using an excel calculator (Retrieved from http://medhealth.leeds.ac.uk/info/2692/research/1826/research/2#pages). A reliable change index of  $\pm$  1.96 was considered a meaningful change over measurement error. Given that Cronbach's alphas cannot be calculated for the LTPA questionnaire, greater than 20 minutes increase of LTPA or MVPA (one bout of LTPA as per the SCI-specific LTPA guidelines for fitness benefits; Martin Ginis et al., 2017) was considered meaningful. The data from the primary and secondary outcomes were also graphed to visually represent individual change among participants in the control and intervention groups. To maintain transparency with the hierarchical multiple regressions originally proposed in our protocol paper, please see online supplemental material (Sweet et al., 2017)

Version Date: 10/19/2017